CLINICAL TRIAL: NCT01197482
Title: Inhaled Steroids and Control of Severe Asthma: Comparison of the AKITA Technology Versus Conventional MDI (INHALE)
Brief Title: Inhaled Steroids and Control of Severe Asthma
Acronym: INHALE
Status: Terminated | Type: Observational
Why Stopped: 6 out of 20 patients were included. The trend towards the treatment of severe asthma has meanwhile developed in a different direction, so that there is no longer any intention to pursue the study objective mentioned here.
Sponsor: University of Giessen (Other)
Collaborators: Activaero GmbH (Industry)
Responsible Party: Principal Investigator, Carmen Brittinger, KKS Sponsor representative, Philipps University Marburg
Other Study IDs: AZ 109/09
Record Dates: First submitted 2010-08-18; First posted 2010-09-09 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Severe Persistent Asthma
Keywords: asthma; inhalation
MeSH Terms: conditions — Asthma; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigational device: AKITA 2 device versus conventional metered-dose inhaler (MDI)

Objectives: To explore if inhalative fluticasone application by means of the AKITA technology would result in a better symptom control in patients with severe persistent asthma as compared to inhalative application of fluticasone by a conventional MDI.

Study design: open label, cross-over (one AKITA, one MDI arm)

Patients: 20 Patients with severe persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* Severe persistent asthma bronchiale with diagnosis according to the criteria of the Global Initiative for Asthma (GINA) executive summary
* Treatment with at least inhaled corticosteroids (ICS) and long acting b agonists (LABA)
* Evidence of inflammatory triggered form of asthma with at least one of the following:
* sensitization to typical aerogenous allergens
* increased Serum IgE levels
* Eosinophilia in peripheral blood
* Proven Eosinophilia in sputum differential (> 3%) in the previous 2 years
* at least 2 exacerbations of asthma within the previous 24 months leading to unscheduled presentation at a health care provider and/or systemic corticosteroid
* Signed informed consent
* Requirements of the local ethics committee are met

Exclusion Criteria:

* Acute exacerbation of asthma within the last 6 weeks Rtot > 350% predicted capillary pO2 < 60mmHG, pCo2 > 50mmHG near fatal asthma or anaphylaxis in history
* Age ≤ 18 and > 80 years
* Active smoking or > 15 pack-years former smoking
* Oral steroid treatment with a prednisolon-equivalent dose exceeding 10 mg per day
* Pregnancy, nursing females
* Female without use of effective contraceptive method
* Treatment with investigational drugs over the past 30 days or during the course of the trial
* Severe and uncontrolled gastroesophageal reflux disease
* Ongoing psychiatric disorder
* Treatment with systemic corticosteroids for any reason other than asthma
* Other active lung diseases
* Medical history of other uncontrolled diseases 3 months prior randomization (e.g. infections, coronary heart diseases and metabolic diseases)
* Any history of malignancy requiring ongoing treatment and/or limiting life-expectancy
* Clinically significant abnormalities in electrocardiogram (ECG) or laboratory exams
* Asthma related to non-steroidal anti-inflammatory drug (NSAID)
* Insulin dependent diabetes mellitus
* Cataract

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe persistent asthma
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Asthma control | 38 weeks
  Changes in asthma control, measured by Juniper Asthma Control Questionnaire during the 16 week treatment period in AKITA versus MDI based steroid application. Physician will assess level of asthma control in accordance with criteria from Gaining Optimal Asthma Control (GOAL) study.

SECONDARY OUTCOMES:
Standardized asthma related quality of life questionnaire (AQLQs) | 38 weeks
  AQLQs will be completed at screening, randomization, crossover and at end of study
Steroid, fluticasone and reliever medication use | 38 weeks
  doses of systemic steroids and fluticasone dosage will be assessed and documented. Frequency of use of reliever medication will be summed from patient's diary and documented.
Lung function | 38 weeks
  Pulmonary function tests (PFT) will be performed and lung function will be assessed by means of spirometry and body plethysmography.
Diffusing capacity for carbon monoxide | 38 weeks
  Diffusing capacity for carbon monoxide will be assessed at rest and holding breath at full inspiration.
Capillary blood gas analysis | 38 weeks
  Capillary blood gas analysis will be obtained from the arterialized ear lobe.
Measurement of Fractional Concentration of Nitric Oxide in Exhaled Air (feNO) | 38 weeks
  feNO will be assessed at each visit. Measurements will be performed following the recommendations of the American Thoracic Society (ATS) and the European Respiratory Society (ERS).
Cell differential in induced sputa | 1 day
  Induced sputum will be obtained at screening if not done within the previous 2 years.
Adrenal function | 38 weeks
  Determination of the fraction of urinary cortisol has been used for screening of adrenal hypo- or hyperfunction and showed to be as effective as 24 hour urinary free cortisol excretion. Urine samples will be obtained at baseline, randomization, crossover and end of study.Values will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Guenther, MD, Principal Investigator — University of Giessen
Locations (3):
- Germany (3):
  - Justus-Liebig-University Giessen, Giessen
  - Lungenfachklinik Waldhof Elgershausen, Greifenstein
  - Philipps-Universität Marburg, Marburg